CLINICAL TRIAL: NCT03315897
Title: Effects of Erythropoietin on Cognitive Functions and Neural Activity in Cognitively Impaired Remitted Patients With Bipolar Disorder or Recurrent Depressive Disorder and Healthy People: Study Protocol for a Randomized, Controlled Trial
Brief Title: Effects of Erythropoietin on Cognition and Neural Activity in Mood Disorders
Acronym: PreTEC-EPO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lars Vedel Kessing (Other)
Collaborators: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other); Lundbeck Foundation (Other)
Responsible Party: Sponsor-Investigator, Lars Vedel Kessing, Professor, MD, DMSc, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Organization: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-16043370; 2016-004023-24 (EudraCT Number); RHP-2017-020 (Other: Danish Data Protection Agency)
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Bipolar Disorder; Cognitive Impairment; Unipolar Depression
Keywords: bipolar disorder; cognition; cognitive dysfunction; erythropoietin; pro-cognitive efficacy; prefrontal cortex; functional magnetic resonance imaging; biomarker; unipolar disorder
MeSH Terms: conditions — Bipolar Disorder; Cognitive Dysfunction; Depressive Disorder | interventions — Erythropoietin; Epoetin Alfa; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erythropoietin (Active Comparator): 12 intravenous infusions of recombinant human erythropoietin (EPO)
  Interventions: Drug: Erythropoietin
- Saline (Placebo Comparator): 12 intravenous infusions of saline (1 ml NaCl)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Erythropoietin — 40.000 IU/ml Erythropoietin (Epoetin alpha; Eprex) diluted with 100 ml saline (0.9% NaCl) is administered 12 times as intravenous infusions over 15 minutes.
  Other Names: Eprex; EPO
  Arms: Erythropoietin
Drug: Saline — 1 ml NaCl is administered 4 times as intravenous infusions over 15 minutes
  Other Names: Placebo
  Arms: Saline

SUMMARY:
The present trial consists of 2 sub-studies that investigate important novel aspects of treatment with erythropoietin (EPO) on cognitive dysfunction in bipolar disorder (BD) and recurrent unipolar depressive disorder (UD) (defined as minimum 2 treatment-requiring depressive episodes). The aims of the trial are three-fold. We aim to investigate the effects of 12 weekly recombinant human EPO infusions on cognition in (i) healthy people with cognitive impairment (substudy 1) and (ii) patients with remitted BD or recurrent UD (substudy 2), and (iii) explore early treatment-associated neural activity changes that may predict subsequent cognitive improvement.

It is hypothesized that:

i. 12 weekly EPO infusions improve cognition in healthy first-degree relatives and remitted BD patients in comparison with saline.

ii. EPO vs. saline-treated participants will display early cognition-related neural activity in the frontal lobes, which will correlate with cognitive improvement.

DETAILED DESCRIPTION:
This trial will include healthy people (sub-study 1) and patients with bipolar disorder or recurrent unipolar depressive disorder in partial or full remission (defined as a score of ≤14 on the Hamilton Depression Rating Scale 17-items and the Young Mania Rating Scale, respectively (sub-study 2) with objectively-verified cognitive dysfunction. Participants will be recruited from Psychiatric Centres in The Mental Health Services in the Capital Region of Denmark, consultant psychiatrists in the Capital Region of Denmark, as well as through advertisements on relevant websites.

The study design comprises 4 major assessments (baseline, week 3, week 13, and a 6 month follow-up after treatment completion) and weekly safety monitoring and study medication infusions during a 12 week treatment period. The baseline assessment is divided into 2 days, 1-3 days apart for practical reasons and to avoid attrition. On the first day of the baseline assessment, participants will perform an fMRI scan. On the second baseline day, participants complete an assessment comprising neuropsychological testing, verbal IQ assessment, and filling in questionnaires concerning subjective cognitive complaints, quality of life, level of functioning, and functional capacity, as well as mood symptom severity ratings. Functional capacity is assessed using a clinician-rated interview and a performance-based task. After 2 weeks of treatment (i.e., 2 doses of EPO or saline) an fMRI scan, neuropsychological testing, mood ratings, and questionnaires on subjective cognitive difficulties are repeated. After treatment completion (week 13) and at the 6 month follow-up, the neuropsychological tests, questionnaires concerning subjective cognitive complaints, quality of life, and functional capacity (self-reported and performance-based) are repeated. Sleep quantity and quality in the past three days is assessed before each of the 4 major assessment time point. Blood samples are collected at baseline, week 3 and 13 for assessment of potential blood-based biomarkers of pro-cognitive effects.

Pharma Consulting Group AB (www.pharmaconsultinggroup.com) has conducted block randomization for each sub-study group, stratified for gender and age (sub-study 1: < or >=30 years; sub-study 2: < or >=35 years). Power calculation was also carried out by Pharma Consulting Group based on findings from a previous RCT in our group assessing the effect of 8 weeks of EPO treatment on the same cognitive composite score. In this trial, the clinically relevant differential change between EPO and saline groups following 12 weeks of treatment is assumed to be at least 0.4 SD (corresponding to a moderate effect size) on the primary outcome with SD of the change of 0.5. Assuming a 10% drop-out rate, we plan to recruit up to n=58 for each sub-study to achieve complete data sets for n=52 participants per sub-study.

Data from the primary, secondary, and tertiary outcomes will be analyzed using Mixed Models Design and Intention to Treat (ITT) analyses. Functional MRI data are pre-processed and analyzed with FMRIB Expert Analysis Tool (FEAT) and the 'randomize' algorithm implemented in FSL (FMRIB Software Library; www.fmrib.ox.ac.uk/fsl). Functional MRI data is analysed using region of interest (ROI) analyses to assess potential differences in neural activity within the dorsal prefrontal cortex and the hippocampi between EPO and placebo groups after 2 weeks of treatment. Exploratory whole-brain analyses are conducted to assess treatment-related activity change in other brain regions. Any differences in neural activity between treatment groups are correlated with potential changes in the primary cognitive composite measure after 2 weeks of treatment (week 3) and after treatment completion (week 13). If this correlation is significant, multiple regression analyses will be performed with adjustment for mood symptoms, age, and gender to assess the potential predictive value of early neural activity change for potential pro-cognitive efficacy after 12 weeks of EPO treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fluent Danish skills and objective cognitive impairment (a total score below cutoff, or scores below cutoff on a minimum of two out of the five subtests (Verbal Learning Test - Immediate, Working Memory Test, Verbal Fluency Test, Verbal Learning Test - Delayed and Processing Speed Test) on the Screen for Cognitive Impairment in Psychiatry - Danish version (SCIP-D).
* Patients must meet the ICD-10 diagnosis of BD (type I and II) or recurrent depressive disorder confirmed using the Schedules for Clinical Assessment in Neuropsychiatry (SCAN) interview.
* Healthy people are eligible even when diagnosed with a less severe mental disorder defined as ICD-10 codes ≥F40.

Exclusion Criteria:

* Schizophrenia or schizoaffective disorder
* Current alcohol or substance misuse disorder (3 months prior to inclusion)
* Daily use of benzodiazepines > 22.5 mg oxazepam
* Diabetes
* Kidney disease
* Renal failure
* Untreated/insufficiently treated arterial hypertension
* Heart diseases (previously diagnosed or abnormal ECG findings during screening)
* Previous serious head trauma
* Neurological illness (including dementia)
* Previous or current epilepsy in patient or first degree family
* Malignancies or thromboses
* Known allergy or antibodies against erythropoietin
* Initial hematocrit > 50% (males) or > 48% (females)
* Initial thrombocyte numbers over normal (>400 billions/L)
* Initial reticulocyte numbers <1‰
* Contraindications against prophylactic thrombosis treatment
* Myeloproliferative disorder, polycythemia
* Pregnancy or breast feeding
* Use of contraceptive medication or other hormonal contraceptives
* Sexually active women in the fertile age, who do not or do not want to use double barrier anticontraceptive methods
* Previous or current history of thromboembolic events or thromboses in patient or first degree family (increased risk of thromboembolic events)
* Overweight (BMI>30) or body weight <45 or >95 kg.
* Previous electroconvulsive therapy (ECT) treatment within last 3 months
* Dyslexia
* Claustrophobia
* Having a pacemaker or other metal implants inside the body
* Reluctance or inability to comply with the protocol requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Cognitive composite score | Change from baseline and week 13
  A cognitive composite based on an average of the Rey Auditory Verbal Learning Test (RAVLT), Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Coding, verbal fluency with the letter "D", WAIS-III Letter-Number Sequencing, Trail Making Test B (TMT B) and Rapid Visual Information Processing (RVP) from Cambridge Cognition (CANTAB).

SECONDARY OUTCOMES:
Rapid Visual Information Processing (RVP) from Cambridge Cognition (CANTAB) | Baseline, two weeks of treatment, week 13, and 6-months follow-up
  Neuropsychological test assessing sustained attention
Functional Assessment Short Test | Baseline, week 13, and 6-months follow-up
  A semi-structured interview assessing level of functioning

OTHER OUTCOMES:
Rey Auditory Verbal Learning Test | Baseline, two weeks of treatment, week 13, and 6-months follow-up
  Neuropsychological test assessing verbal memory
Trail Making Test Part A | Baseline, two weeks of treatment, week 13, and 6-months follow-up
  Neuropsychological test assessing attention and processing speed
Trail Making Test Part B | Baseline, two weeks of treatment, week 13, and 6-months follow-up
  Neuropsychological test assessing executive functions
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Coding | Baseline, two weeks of treatment, week 13, and 6-months follow-up
  Neuropsychological test assessing attention
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Digit Span | Baseline, two weeks of treatment, week 13, and 6-months follow-up
  Neuropsychological test assessing executive functions
WAIS-III Letter-Number Sequencing | Baseline, two weeks of treatment, week 13, and 6-months follow-up
  Neuropsychological test assessing executive functions
Verbal fluency with the letter "D" and 'S" | Baseline, two weeks of treatment, week 13, and 6-months follow-up
  Neuropsychological test assessing executive functions
One Touch Stockings of Cambridge | Baseline, two weeks of treatment, week 13, and 6-months follow-up
  A computerized neuropsychological test assessing executive functions
Spatial Working Memory (SWM) from Cambridge Cognition | Baseline, two weeks of treatment, week 13, and 6-months follow-up
  Neuropsychological test assessing sustained attention
Brief University of California, San Diego Performance-Based Skills Assessment-B | Baseline, week 13, and 6-months follow-up
  Objective, performance-based assessment of level of functioning
Sheehan Disability Scale | Baseline, week 13, and 6-months follow-up
  Visual analogue scale assessing level of functioning (i.e., the magnitude to which social, professional, and everyday life is impaired by symptoms). Each of the three subscale items have numerical scores that range from 0 to 10 with higher scores representing worse outcomes. These subscale items can be summed into a total dimensional measure reflecting global functional impairment with scores that range from 0 (no functional impairment at all) to 30 (severe functional impairment).
The Assessment of Quality of Life | Baseline, week 13, and 6-months follow-up
  Questionnaire on quality of life
World Health Organization Quality of Life | Baseline, week 13, and 6-months follow-up
  Questionnaire on quality of life
Cognitive Complaints in Bipolar Disorder Rating Assessment | Baseline, week 13, and 6-months follow-up
  Questionnaire on subjective cognitive complaints
Work and Social Adjustment Scale | Baseline, week 13, and 6-months follow-up
  Questionnaire on occupational functioning (work and social adjustment). The questionnaire consists of five subscale items with numerical scores that range from 0 (reflecting no impairment at all) to 8 (reflecting severe impairment). These subscale items can be summed into a total dimensional measure assessing global work and social adjustment with scores that range from 0 to 40 (with higher scores reflecting worse outcomes).

CONTACTS AND LOCATIONS:
Overall Officials: Lars V. Kessing, Prof., Principal Investigator — Mental Health Services, Capital Region of Denmark, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark, 2100; Kamilla W. Miskowiak, Prof., Study Director — Mental Health Services, Capital Region of Denmark, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark, 2100
Locations (1):
- Mental Health Services, Capital Region of Denmark, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Macoveanu J, Petersen JZ, Mariegaard J, Jespersen AE, Cramer K, Bruun CF, Madsen HO, Jorgensen MB, Vinberg M, Fisher PM, Knudsen GM, Hageman I, Ehrenreich H, Kessing LV, Miskowiak KW. Effects of erythropoietin on cognitive impairment and prefrontal cortex activity across affective disorders: A randomized, double-blinded, placebo-controlled trial. J Psychopharmacol. 2024 Apr;38(4):362-374. doi: 10.1177/02698811241237869. Epub 2024 Mar 22. PMID 38519416
- [Derived] Petersen JZ, Schmidt LS, Vinberg M, Jorgensen MB, Hageman I, Ehrenreich H, Knudsen GM, Kessing LV, Miskowiak KW. Effects of recombinant human erythropoietin on cognition and neural activity in remitted patients with mood disorders and first-degree relatives of patients with psychiatric disorders: a study protocol for a randomized controlled trial. Trials. 2018 Nov 6;19(1):611. doi: 10.1186/s13063-018-2995-7. PMID 30400939